CLINICAL TRIAL: NCT05755776
Title: To Evaluate the Efficacy and Safety of Tenofovir Amibufenamide in Chronic Hepatitis B (CHB) Patients With Low-level Viraemia (LLV) After Entecavir Treatment
Brief Title: The Efficacy and Safety of Tenofovir Amibufenamide to Treat Low-level Viraemia After Entecavir Treatment
Acronym: POWER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-10234-A005
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-10

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis b; Entecavir; Tenofovir Amibufenamide; Low-level viraemia
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ETV group: Participants in this group will continue ETV daily until the end of the study.
- TMF group: Participants in this group will switch to TMF 25 mg, daily until the end of the study.
  Interventions: Drug: TMF

INTERVENTIONS:
Drug: TMF — switch ETV to TMF
  Other Names: Heng Mu
  Groups: TMF group

SUMMARY:
The goal of this observational study is to explore the efficacy and safety of Tenofovir Amibufenamide (TMF) in Entecavir (ETV) treated chronic hepatitis B patients with low-level viraemia. The main question it aims to answer is:

* The efficacy and safety of TMF in chronic hepatitis B patients with low-level viraemia.
* What is the appropriate treatment for ETV treated chronic hepatitis B patients with low-level viraemia.

Participants will choose to maintain their original regimen (ETV) or switch to TMF After being fully informed of the benefits and risks of treatment.

Researchers will compare ETV and TMF to see if there is a difference in the efficacy of the two drugs in chronic hepatitis B patients with low-level viraemia.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and sign a written informed consent, which must be obtained prior to screening.
2. Male and non-pregnant, non-lactating female subjects who have reached the age of 18-65 years (based on the date of signed informed consent). Female subjects of childbearing age with a negative serum pregnancy test.
3. Documented signs of chronic HBV infection (e.g., HBsAg positive for more than 6 months.
4. Subjects treated with ETV over 1 year will be able to be enrolled in the study.
5. Subjects with 20 ≤ HBV-DNA < 2000 IU/mL at screening (including intermittent and continuous low-level viraeima).
6. Must be willing and able to comply with all study requirements.

Exclusion Criteria:

1. Female patients who are pregnant or breastfeeding or who plan to become pregnant during the study period.
2. Men and women of childbearing potential who are unwilling to use an "effective" method of contraception as defined in the protocol during the study period.
3. Co-infection with HAV HCV, HIV, HDV or HEV; or co-infection with autologous liver, metabolism-related fatty liver, or drug-induced liver injury.
4. Diagnosis of hepatocellular carcinoma by imaging (with evidence of hepatocellular carcinoma)
5. Patients who have received a solid organ or bone marrow transplant
6. History of malignancy within 5 years prior to screening, except for specific tumors cured by surgical resection (basal cell dermal skin cancer, etc.); patients evaluated for probable malignancy were ineligible.
7. Currently receiving treatment with immunomodulators (e.g., corticosteroids), investigational drugs, nephrotoxic drugs, or drugs capable of regulating renal excretion. Drugs that modulate renal excretion.
8. Renal, cardiovascular, pulmonary, or neurological disease that is considered severe by the investigator.
9. Severe bone disease (e.g., osteochondrosis, chronic osteomyelitis, osteogenesis imperfecta, chondromalacia) or multiple fractures.
10. Subjects receiving a contraindicated combination drug (subjects receiving a contraindicated drug require a minimum 30-day washout period) and known hypersensitivity reactions to study drugs, metabolites or formulation excipients.
11. Current alcohol or drug abuse that, in the investigator's judgment, may interfere with the subject's compliance with study requirements.
12. Any other clinical condition that, in the opinion of the investigator, would render the subject unsuitable for the study or unable to comply with the dosing requirements medical condition or prior treatment.
13. Prior or existing clinical liver failure (Child-Pugh score ≥ grade B).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population was chronic hepatitis B patients with LLV (HBV DNA from 20-to 2000IU/mL) of ETV treatment from multiple centers across mainland China.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The proportions of undetectable HBV DNA in patients treated with ETV and TMF at week 48. | 48 weeks
  Undetectable HBV DNA is defined as below 20 IU/mL.

SECONDARY OUTCOMES:
The proportions of undetectable HBV DNA in patients treated with ETV and TMF at week 24. | 24 weeks
  Undetectable HBV DNA is defined as below 20 IU/mL.
The proportions of ALT normalization in patients treated with ETV and TMF at week 24 and 48. | 24 weeks and 48 weeks
  There are two criteria for ALT normalization. Criteria1: below 40 U/L. Criteria2: Males: ALT<30U/L, female: ALT<19U/L.
Comparing pgRNA levels from baseline at week 24 and 48. | 24 weeks and 48 weeks
Comparing HBcrAg levels from baseline at week 24 and 48. | 24 weeks and 48 weeks
The proportions of undetectable pgRNA in patients treated with ETV and TMF at week 24 and 48. | 24 weeks and 48 weeks
  Undetectable pgRNA is defined as below 100 pg/mL.
The proportions of undetectable HBcrAg in patients treated with ETV and TMF at week 24 and 48. | 24 weeks and 48 weeks
Comparing degree of liver fibrosis from baseline at week 24 and 48. | 24 weeks and 48 weeks
  Evaluation of liver fibrosis including Fibroscan, APRI and FIB-4.
Comparing the change of creatinine clearance rate from baseline at week 24 and 48. | 24 weeks and 48 weeks
The types, incidence and severity of adverse events and serious adverse events during treatment were evaluated in both groups | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Peng Hu, phD, Study Director — The Second Affiliated Hospital of Chongqing Medical University
Locations (13):
- China (13):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Central Hospital, Chongqing
  - Affiliated Hospital of Guangxi Medical University, Guangxi
  - Hepatobiliary disease of Jilin Province, Jilin
  - The First People's Hospital of Yunnan Province, Kunming
  - the Second People's Hospital of Yunnan Province, Kunming
  - Nanjing Second Hospital, Nanjing
  - The Second Hospital of Ningbo, Ningbo
  - Shanghai East Hospital, Shanghai
  - Shuguang Hospital, Shanghai, China., Shanghai
  - The Sixth People's Hospital of Shenyang, Shenyang
  - The First People's Hospital of Taicang, Taicang
  - The Fourth People's Hospital of Zibo, Zibo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu J, Liang W, Jing W, Liu M. Countdown to 2030: eliminating hepatitis B disease, China. Bull World Health Organ. 2019 Mar 1;97(3):230-238. doi: 10.2471/BLT.18.219469. Epub 2019 Jan 28. PMID 30992636
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] Sun Y, Wu X, Zhou J, Meng T, Wang B, Chen S, Liu H, Wang T, Zhao X, Wu S, Kong Y, Ou X, Wee A, Theise ND, Qiu C, Zhang W, Lu F, Jia J, You H. Persistent Low Level of Hepatitis B Virus Promotes Fibrosis Progression During Therapy. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2582-2591.e6. doi: 10.1016/j.cgh.2020.03.001. Epub 2020 Mar 6. PMID 32147592
- [Background] Kim JH, Sinn DH, Kang W, Gwak GY, Paik YH, Choi MS, Lee JH, Koh KC, Paik SW. Low-level viremia and the increased risk of hepatocellular carcinoma in patients receiving entecavir treatment. Hepatology. 2017 Aug;66(2):335-343. doi: 10.1002/hep.28916. Epub 2016 Dec 24. PMID 28012257
- [Background] Wang J, Sheng Q, Ding Y, Chen R, Sun X, Chen X, Dou X, Lu F. HBV RNA virion-like particles produced under nucleos(t)ide analogues treatment are mainly replication-deficient. J Hepatol. 2018 Apr;68(4):847-849. doi: 10.1016/j.jhep.2017.10.030. Epub 2017 Nov 4. No abstract available. PMID 29113914
- [Background] Yuen MF, Seto WK, Fung J, Wong DK, Yuen JC, Lai CL. Three years of continuous entecavir therapy in treatment-naive chronic hepatitis B patients: VIRAL suppression, viral resistance, and clinical safety. Am J Gastroenterol. 2011 Jul;106(7):1264-71. doi: 10.1038/ajg.2011.45. Epub 2011 Mar 1. PMID 21364549
- [Background] Korean Association for the Study of the Liver (KASL). KASL clinical practice guidelines for management of chronic hepatitis B. Clin Mol Hepatol. 2019 Jun;25(2):93-159. doi: 10.3350/cmh.2019.1002. Epub 2019 Jun 12. No abstract available. PMID 31185710
- [Background] Ogawa E, Nomura H, Nakamuta M, Furusyo N, Koyanagi T, Dohmen K, Ooho A, Satoh T, Kawano A, Kajiwara E, Takahashi K, Azuma K, Kato M, Shimoda S, Hayashi J; Kyushu University Liver Disease Study (KULDS) Group. Tenofovir alafenamide after switching from entecavir or nucleos(t)ide combination therapy for patients with chronic hepatitis B. Liver Int. 2020 Jul;40(7):1578-1589. doi: 10.1111/liv.14482. Epub 2020 Apr 30. PMID 32304611
- [Background] Liu Z, Jin Q, Zhang Y, Gong G, Wu G, Yao L, Wen X, Gao Z, Huang Y, Yang D, Chen E, Mao Q, Lin S, Shang J, Gong H, Zhong L, Yin H, Wang F, Hu P, Xiao L, Li C, Wu Q, Sun C, Niu J, Hou J; TMF Study Group. Randomised clinical trial: 48 weeks of treatment with tenofovir amibufenamide versus tenofovir disoproxil fumarate for patients with chronic hepatitis B. Aliment Pharmacol Ther. 2021 Nov;54(9):1134-1149. doi: 10.1111/apt.16611. Epub 2021 Sep 29. PMID 34587302